CLINICAL TRIAL: NCT03659071
Title: Hematopoietic Stem Cell Transplantation and Childhood Leukemia: Quality of Life in SIbling DONors, Years After the Donation
Brief Title: Hematopoietic Stem Cell Transplantation and Childhood Leukemia Quality of Life in SIbling DONors
Acronym: SIDONY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCAPHM17_0169
Record Dates: First submitted 2018-08-17; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Hematopoietic/Lymphoid Cancer
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DONORS (Experimental): donors from the siblings of survivors of acute childhood leukemia who have received hematopoietic stem cell transplantation questionnaire VSP-A will be performed
  Interventions: Other: questionnaire VSP-A
- NON DONORS (Other): non-donor siblings. questionnaire VSP-A will be performed
  Interventions: Other: questionnaire VSP-A

INTERVENTIONS:
Other: questionnaire VSP-A — VSP-A (écu et Santé Perçue de l'Adolescent et de l'enfant): Lived and perceived health of the adolescent and child developed from the exclusive point of view of the child, for which reference values in French population are available. The self-questionnaire used is a questionnaire developed and validated in French for children and adolescents, according to the standards in force, apprehending 9 dimensions (vitality, psychological well-being, relations with friends, leisure, family relations, good physical, relationships with teachers, school work, self-esteem)

SUMMARY:
The childhood cancer experience necessarily impacts the entire family. In this context, particular attention should be paid to the donor siblings of hematopoietic stem cells in the context of treatment of leukemia by grafting.

The results of the little existing work on the long-term fate of stem cell donor siblings of cancer survivors report psychosocial consequences, particularly for real post-traumatic stress in distant siblings.

Few studies have explored the medium and long-term impact of the disease, as well as donation, on a broader set of domains structuring the quality of life, through validated quantitative tools.

In France, since 2004, the LEA program (Leukemia of the Child and Adolescent) aims to assess the determinants of the state of health and quality of life in the medium and long term, patients treated for acute childhood leukemia after 1980.

The main objective of this study is to evaluate, at a distance from the transplant, the quality of life of donors from the siblings of survivors of acute childhood leukemia who received a hematopoietic stem cell transplant compared with non-donor siblings.

The SIDONY ancillary study will be proposed to families of LEA patients who have received a geno-identical sibling haematopoietic stem cell transplant (population of interest) and to families whose LEA patient has not been treated by sibling transplantation. geno-identical but still declaring to have siblings (main comparator group). Each family will be contacted by mail and the management of inclusions will be managed by the Epidemiology and Health Economics Department of AP-HM (Marseille).

Information not routinely available in the LEA database will be collected from the siblings (self-questionnaire, in addition, for each surviving child included in the cohort, data are available: sociodemographic; characteristics of the initial disease and therapeutic received; physical sequelae; quality of life.

The population meeting the inclusion criteria represents 2639 subjects: 337 donors and 2302 non-donors, making it possible to obtain high powers for analyzes (linear regression, multilevel analyzes, etc.). This study could identify profiles of siblings for whom the quality of life seems particularly impaired, potential object of individual interventions (remediation ...).

DETAILED DESCRIPTION:
The childhood cancer experience necessarily impacts the entire family. In this context, particular attention should be paid to the donor siblings of hematopoietic stem cells in the context of treatment of leukemia by grafting.

The results of the little existing work on the long-term fate of stem cell donor siblings of cancer survivors report psychosocial consequences, particularly for real post-traumatic stress in distant siblings. disease. Few studies have explored the medium and long-term impact of the disease, as well as donation, on a broader set of domains structuring the quality of life, through validated quantitative tools.

In France, since 2004, the LEA program (Leukemia of the Child and Adolescent) aims to assess the determinants (medical, socio-economic, behavioral and environmental) of the state of health and quality of life in the medium and long term, patients treated for acute childhood leukemia after 1980. To document the quality of life of their self-reported hematopoietic stem cell donor siblings and their perception of the impact that experience of cancer in the family has had on their medium and long-term future, the organization of the LEA program can easily be extended to the establishment of an ancillary study.

objectives The main objective of this study is to evaluate, at a distance from the transplant, the quality of life of donors from the siblings of survivors of acute childhood leukemia who received a hematopoietic stem cell transplant compared with non-donor siblings.

The secondary objectives are: (a) to compare the quality of life of siblings with that of the general population; (b) to compare the quality of life of the siblings with that of the surviving patients; (c) to identify the determinants (demographic, socioeconomic, family and history of cancer) of the medium-long-term quality of life of this family; (d) remotely evaluate the donation's use of the donor sire care system as a tracer of the impact of the donation; (e) remotely evaluate the gift of the social integration of the donor sibship, particularly in terms of schooling.

The SIDONY ancillary study will be proposed to families of LEA patients who have received a geno-identical sibling haematopoietic stem cell transplant (population of interest) and to families whose LEA patient has not been treated by sibling transplantation. geno-identical but still declaring to have siblings (main comparator group). Each family will be contacted by mail and the management of inclusions will be managed by the Epidemiology and Health Economics Department of AP-HM (Marseille).

Information not routinely available in the LEA database will be collected from the siblings (self-questionnaire, to be returned by post): sociodemographic and socio-economic data relating to the siblings and the family; data concerning the quality of life of the siblings; psycho-behavioral and cognitive data; data on the state of health of the siblings; social inclusion data; recourse to the health care system. In addition, for each surviving child included in the cohort, data are available: sociodemographic; characteristics of the initial disease and therapeutic received; physical sequelae; quality of life.

Feasibility and practical impact The population meeting the inclusion criteria represents 2639 subjects: 337 donors and 2302 non-donors, making it possible to obtain high powers for analyzes (linear regression, multilevel analyzes, etc.). This study could identify profiles of siblings for whom the quality of life seems particularly impaired, potential object of individual interventions (remediation ...).

ELIGIBILITY:
Inclusion Criteria:

1. experimental group familly:

   * child included in the LEA cohort
   * having received allogeneic treatment of geno-identical sibling haematopoietic stem cells
2. Criteria for the inclusion of siblings (experimental group)

   * be the brother (or sister) donor of hematopoietic stem cells
   * currently at least 8 years old
   * give consent to participate in the study
   * be allowed to participate in the study by his parents or legal representatives
3. Control group familly

   * child included in the LEA cohort
   * who did not benefit from allogeneic hematopoietic stem cell transplantation of geno-identical siblings
   * and declaring having a sibling
4. Criteria for the inclusion of siblings (control group)

   * currently at least 8 years old
   * to be the closest brother (or sister) in the LEA patient's age (in the case of multiple siblings)
   * give consent to participate in the study
   * be allowed to participate in the study by his parents or legal representatives In order to respect the balance within the family, a questionnaire may be distributed to other brothers and sisters who claim it.

Exclusion Criteria:

not to be allowed to participate in the study by his parents or legal representatives

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1187 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Quality of life scores | 1 day
  VSPA questionnaire score
  Each item is rated from 1 to 5, depending on the answer:
  * Never / not at all,
  * arement / a little
  * sometimes / medium
  * some / many
  * Always enormously The scores were calculated according to the algorithm defined by the author of the questionnaire: the score of each dimension was obtained from the average of the answers given for the items of the dimension concerned.
  Scores range from 0 (the worst quality of life) to 100 (the best).

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France